CLINICAL TRIAL: NCT01403831
Title: Trial to Examine Text-message Based mHealth in Emergency Department Patients With Diabetes
Acronym: TExT-MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sanjay Arora, PI, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-11-00084; Mobilizing for Health (Other Grant/Funding Number: McKesson Foundation)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text messages (Experimental): Patients randomized to this arm will receive daily text messages to their mobile phones consisting of educational materials, motivational materials, trivia questions, and challenges to engage in healthy lifestyle choices
  Interventions: Other: Daily text messages
- Control (No Intervention)

INTERVENTIONS:
Other: Daily text messages — 2-3 times daily text messages regarding diabetes care and healthy lifestyle choices
  Arms: Text messages

SUMMARY:
The investigators propose an innovative, ED-based mHealth intervention: TExT-MED (Trial to Examine Text-Based mHealth for Emergency department patients with Diabetes). TExT-MED is a technologically simple solution using unidirectional daily text messages to consisting of educational materials, trivia questions and challenges promoting healthy lifestyle choices and reminders to check blood sugar, take medications and go to clinic appointments. The investigators believe TExT-MED will improve health outcomes including blood glucose control and encourage weight loss, healthy eating and exercise. TExT-MED is low cost, easy to use and can be quickly adapted to other practice environments.

ELIGIBILITY:
Inclusion Criteria:

1) ≥18 years old 2) have Type 2 diabetes 3) have a text message capable mobile phone 4) know how to receive text messages 5) speak and read English or Spanish and 6) have a HbA1C ≥8%.

Exclusion Criteria:

1) overt psychosis 2) unable to provide informed consent and 3) pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C at 6 months | 6 months

SECONDARY OUTCOMES:
DIet/ Weight Loss | 6 months
Diabetes self-efficacy/empowerment | 6 months
Diabetes knowledge | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Arora S, Peters AL, Agy C, Menchine M. A mobile health intervention for inner city patients with poorly controlled diabetes: proof-of-concept of the TExT-MED program. Diabetes Technol Ther. 2012 Jun;14(6):492-6. doi: 10.1089/dia.2011.0252. Epub 2012 Apr 23. PMID 22524591